CLINICAL TRIAL: NCT04468893
Title: Effectiveness of a Self-applied Positive Psychology Online Intervention Program "Mental Health COVID-19" in Mexican Population: A Randomized Controlled Trial.
Brief Title: Online Positive Psychology Intervention for Depression and Anxiety Due to COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Internacional de Valencia (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); Universidad Autonoma de Ciudad Juarez (Other)
Responsible Party: Principal Investigator, Alejandro Domínguez Rodríguez, External professor, Universidad Internacional de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIU-PP
Record Dates: First submitted 2020-07-10; First posted 2020-07-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Anxiety; Depression; Sleep Disturbance
MeSH Terms: conditions — Anxiety Disorders; Depression; Parasomnias

STUDY DESIGN:
Intervention Model Description: The study has two arms, one is the intervention group that receives the treatment in addition to a chat service and the other is the comparison group that will receive treatment without the chat service. The patients in both groups will be evaluated pre and post/treatment. The participants are assigned randomly to the intervention or comparison group.
Who Masked: Participant
Masking Description: The patients are not aware that there is an intervention group and a comparison group, the participants are not related and do not know each other. The conditions of the study are only known by the researcher, the therapists, and the Ethics Committee of ELPAC-UU Universidad de Ciencias del Comportamiento
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology Intervention with chat (Experimental): Participants in this group will receive from 15 sessions of a Positive Psychology focused on the increase of wellbeing and sleep quality and decrease of anxiety and depression with the support of a chat service provided by therapists.
  Interventions: Behavioral: Online Intervention Mental Health COVID-19
- Positive Psychology Intervention without chat (Active Comparator): Participants in this group will receive from 15 sessions of a Positive Psychology focused on the increase of wellbeing and sleep quality and decrease of anxiety and depression without the support of the chat service.
  Interventions: Behavioral: Online Intervention Mental Health COVID-19

INTERVENTIONS:
Behavioral: Online Intervention Mental Health COVID-19 — The Online Intervention Mental Health COVID-19 aims to provide to the target population a self-applied intervention based primarily on Positive Psychology, aimed at the recognition and development of strengths and virtues from the well-being approach. In addition, it is supported by elements of Cognitive Behavioral Therapy such as the components of emotion and the Antecedent-Response-Consequence (ARC) model of emotions. Elements of Behavioral Activation Therapy are also included, such as the importance of physical exercise and the relationship between physical anxiety and its effects on anxiety and depression. The intervention is made up of 15 modules that are adapted to the symptoms that the population may suffer from the global contingency caused by the COVID-19 pandemic. In addition to the Positive Psychology modules, a module with psychoeducation on grief and loss was added.

SUMMARY:
This study evaluates the effectiveness of a Positive Psychology intervention, that is focused on increasing the positive emotions and strengths of human beings. It is compared to the effectiveness of an online treatment with the change of the same participants before and after receiving the treatment accompanied by a chat support service vs. the treatment solely. The changes are being assessed through worldwide validated measures such as psychometrics.

DETAILED DESCRIPTION:
The outbreak of the new coronavirus 2019 (COVID-19) has become a public health emergency of international concern that has not only threatened people's physical health but has also affected mental health and psychological well-being. Among the several symptoms can be observed an affected sleep quality, symptoms of posttraumatic stress disorder, anxiety, depression, and complicated grief, among others.

To provide treatment in such conditions where face-to-face sessions are not possible, and the number of patients surpasses the number of available therapists it will be implemented an online intervention based on positive psychology. positive Psychology has been defined as the scientific study of positive experiences, positive individual traits, the institutions that facilitate their development, and the programs that help to improve the quality of life of the individuals while preventing or reducing the incidence of psychopathology.

The online intervention system Mental Health Platform COVID-19 will be delivered in 15 modules interconnected, implemented one per session. The objective of this study is to assess the efficacy and moderators of change of an intervention program based on the Positive Psychology approach for the reduction of anxious and depressive symptoms, increase of positive emotions and sleep quality during and after the contingency by COVID-19 by means of a telepsychology.

This study will have two intervention groups, one that will receive the online intervention plus a chat added element. The chat service will be provided by clinical therapists through the Tawk application where participants can receive help if they have questions about a module and its activities or a technical problem, in addition to other functions. The comparison group will receive the same intervention however will not include the chat service. In both conditions, the participants will be measured pre and post. The subjective measures will include the following psychometrics:

1. Scale of Post-traumatic Stress Traits in the Mexican Youth Exposed to Social Violence.
2. Widespread fear Scale.
3. State-Trait Anxiety Inventory (STAI).
4. Generalized Anxiety Disorder 7-item (GAD-7) scale.
5. Beck Depression Scale (BDI-II)
6. The Pittsburgh Sleep Quality Index
7. Suicidal Thoughts Scale.

ELIGIBILITY:
Inclusion Criteria:

* To have access to a communication device with access to the internet (computer, tablet, and mobile).
* To have a valid email address.
* To have basic digital skills in the use of an operational system and internet browsing.
* To understand Spanish since all the contents are in this language

Exclusion Criteria:

* To have a diagnosis of psychotic disorder.
* To be receiving psychological and / or pharmacological treatment during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Decrease in the score of Anxiety symptoms | [Time Frame: 2 weeks to one month, depending on the development of the patient and the completion of the 15 modules.]
  The State/Trait Anxiety Inventory consists of two subscales of 20 items each that measure anxiety as a transient state of tension (Scale A-State), and as a characteristic of the personality relatively stable over time (Scale B -trait). The items are composed by an assertion to which the subject responds indicating their degree of identification. In the case of state anxiety, the scale goes from 1 (not at all), 2 (somewhat), 3 (moderately), 4 (very much), while in the trait anxiety it ranges from 1 (almost never), 2 (sometimes), 3 (often), 4 (almost always). In both, a percentage of the items evaluate well-being or absence of anxiety, while the rest of the items to the presence of anxiety. Scores range from 20 to 80, in each subscale, with higher scores correlating with greater anxiety. It is expected a statistically significant decrease (P < 0.05) in the anxiety symptoms.
Change in the symptoms of depression | [Time Frame: 2 weeks to one month, depending on the development of the patient and the completion of the 15 modules.]
  The Beck Depression Inventory is a self-report that provides a measure of the presence and severity of depression. Contains 21 items indicative of symptoms such as sadness, crying, loss of pleasure, feelings of failure and guilt, suicidal thoughts or desires, pessimism, etc. Each item is answered on a 4-point scale, from 0 to 3, where each number is identified differently for each item, in all of them 0 means absence and 3 full presence (e.g. sadness), except for items 16 (changes in the sleep pattern) and 18 (changes in appetite) that contain 7 categories. The minimum and maximum scores in the test are 0 and 63. Cut-off points ha that allow classifying those evaluated in one of the following four groups: 0-13, minimum depression; 14-19, mild depression; 20-28, moderate depression; and 29-63, severe depression. It is expected a statistically significant decrease (P < 0.05) in the depression symptoms.
Change in the symptoms of General Anxiety Disorder | [Time Frame: 2 weeks to one month, depending on the development of the patient and the completion of the 15 modules.]
  On the Generalized Anxiety Disorder 7-item (GAD-7) scale subjects are asked how often, during the last 2 weeks, they have been bothered by each of the 7 core symptoms of generalized anxiety disorder. Response options are "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively. Therefore, GAD-7 scores range from 0 to 21, with scores of ≥5, ≥10, and ≥15 represent mild, moderate, and severe anxiety symptom levels, respectively. It is expected a statistically significant decrease (P < 0.05) in the General Anxiety symptoms.
Change in the score of Posttraumatic stress symptoms | [Time Frame: 2 weeks to one month, depending on the development of the patient and the completion of the 15 modules.]
  The Scale of Post-traumatic Stress Traits in the Mexican Youth Exposed to Social Violence It is a brief scale with 24 symptoms corresponding to the diagnosis of PTSD, to respond by self-report, and a scale was used discretely from 1 (strongly disagree) to 4 (strongly agree). The total score was obtained by arithmetic sum. The minimum possible is 24 and the maximum 96. It is expected a statistically significant decrease (P < 0.05) in the posttraumatic stress symptoms.
Changes in the Widespread fear Scale | [Time Frame: 2 weeks to one month, depending on the development of the patient and the completion of the 15 modules.]
  It is composed of seven items with options of 0 = nothing, 3 = a lot, and measures the fear in its emotional component, that is, the fear to adversities in the context and the feelings it disseminates, as well as others economic and social fears, in this case, adapted for the Sars-Cov2 pandemic. In previous studies, an acceptable internal consistency of .95 was reached. It consists of several items about the fear of being a SARS Cov2 victim in diverse contexts. In the present study, a Cronbach alpha coefficient of 0.96 was obtained. It is expected a statistically significant decrease (P < 0.05) in the widespread fear symptoms.
Change in the score of The Pittsburgh Sleep Quality Index. | [Time Frame: 2 weeks to one month, depending on the development of the patient and the completion of the 15 modules.]
  This instrument assesses the quality patterns of sleep. It differentiates the "poor" and "good" sleep by measuring seven areas, where the range score of answers are from 0 to 3, the global sum of this scale can be a value between 0 to 60, and the cutoff point is "5" that indicates a "poor" sleep quality. It is expected a statistically significant increase (P < 0.05) in the Sleep Quality Index.

SECONDARY OUTCOMES:
Change on the Suicidal Thoughts Scale | [Time Frame: 2 weeks to one month, depending on the development of the patient and the completion of the 15 modules.]
  This scale aims to assess the frequency of attitudes, behaviors and plans to commit suicide. It is divided into 19 items with a response option of 0 to 2, giving a total of 0 to 38 where a score equal to or greater than 10 indicates an existing risk of suicide. This scale has been validated in the Mexican population (González-Macip & Díaz-Martínez, 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Anabel de la Rosa Gómez, PhD, Study Chair — Universidad Nacional Autonoma de Mexico; Paulina Arenas Landgrave, PhD, Study Chair — Universidad Nacional Autonoma de Mexico; Jasshel Teresa Salinas-Saldivar, MD, Study Chair — Universidad Autónoma de Ciudad Juárez; Flor Rocio Ramirez-Martinez, PhD, Study Chair — Universidad Autónoma de Ciudad Juárez; Sofía Cristina Martínez Luna, MD, Study Chair — Universidad Nacional Autonoma de Mexico
Locations (1):
- Universidad Autónoma de Ciudad Juárez, Juárez, Chihuahua, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a server of the journal(s) that we will publish the articles that will be the result of this study. The protocol of the study is currently in progress to be published, in this article will be included such study protocol, the informed consent is already shared in the register of clinical trials.
Supporting Information: Study Protocol, ICF
Time Frame: This data will be available approximately in december 2020 and it will be permanently available. It will be shared in the databases of the journal where the article(s) will be published
Access Criteria: Through the servers of the journal(s) where we will publish the articles.

REFERENCES:
- [Background] Davies EB, Morriss R, Glazebrook C. Computer-delivered and web-based interventions to improve depression, anxiety, and psychological well-being of university students: a systematic review and meta-analysis. J Med Internet Res. 2014 May 16;16(5):e130. doi: 10.2196/jmir.3142. PMID 24836465
- [Background] Chávez-Valdez SM, Esparza-Del Villar OA, Ríos Velasco-Moreno L. Validation of a Scale of Post-traumatic Stress Traits in the Mexican Youth Exposed to Social Violence. Journal of Aggression, Maltreatment & Trauma [Internet]. Informa UK Limited; 2020 Jan 8;1-13. DOI: http://dx.doi.org/10.1080/10926771.2019.1710635
- [Background] Wang C, Pan R, Wan X, Tan Y, Xu L, Ho CS, Ho RC. Immediate Psychological Responses and Associated Factors during the Initial Stage of the 2019 Coronavirus Disease (COVID-19) Epidemic among the General Population in China. Int J Environ Res Public Health. 2020 Mar 6;17(5):1729. doi: 10.3390/ijerph17051729. PMID 32155789
- [Background] Beck AT, Steer, RA, Brown, GK. Manual for Beck Depression Inventory-II. (1996) San Antonio, TX: Psychological Corporation.
- [Result] Beck AT, Steer RA, Ranieri WF. Scale for Suicide Ideation: psychometric properties of a self-report version. J Clin Psychol. 1988 Jul;44(4):499-505. doi: 10.1002/1097-4679(198807)44:43.0.co;2-6. PMID 3170753
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Hishinuma ES, Miyamoto RH, Nishimura ST, Nahulu LB, Andrade NN, Makini GK Jr, Yuen NY, Johnson RC, Kim SP, Goebert DA, Guerrero AP. Psychometric properties of the state-trait anxiety inventory for Asian/Pacific-islander adolescents. Assessment. 2000 Mar;7(1):17-36. doi: 10.1177/107319110000700102. PMID 10668003
- [Result] Walsh S, Szymczynska P, Taylor SJC, Priebe S. The acceptability of an online intervention using positive psychology for depression: A qualitative study. Internet Interv. 2018 Jul 8;13:60-66. doi: 10.1016/j.invent.2018.07.003. eCollection 2018 Sep. PMID 30206520
- [Result] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Derived] Dominguez-Rodriguez A, Sanz-Gomez S, Gonzalez Ramirez LP, Herdoiza-Arroyo PE, Trevino Garcia LE, de la Rosa-Gomez A, Gonzalez-Cantero JO, Macias-Aguinaga V, Arenas Landgrave P, Chavez-Valdez SM. Evaluation and Future Challenges in a Self-Guided Web-Based Intervention With and Without Chat Support for Depression and Anxiety Symptoms During the COVID-19 Pandemic: Randomized Controlled Trial. JMIR Form Res. 2024 Sep 30;8:e53767. doi: 10.2196/53767. PMID 39348893
- [Derived] Dominguez-Rodriguez A, De La Rosa-Gomez A, Hernandez Jimenez MJ, Arenas-Landgrave P, Martinez-Luna SC, Alvarez Silva J, Garcia Hernandez JE, Arzola-Sanchez C, Acosta Guzman V. A Self-Administered Multicomponent Web-Based Mental Health Intervention for the Mexican Population During the COVID-19 Pandemic: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Nov 16;9(11):e23117. doi: 10.2196/23117. PMID 33196449

DOCUMENTS (1):
  • Informed Consent Form (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT04468893/ICF_000.pdf